CLINICAL TRIAL: NCT05037747
Title: Effects of Time-restricted Feeding on Obese Patients With Chronic Kidney Disease Stage 3-4: a Pilot Study
Brief Title: Effects of TRF on Obese Patients With CKD Stage 3-4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Liu Xu-sheng, Head of Nephrology, Director, Principal Investigator, Clinical Professor, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YF2021-142
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Time Restricted Feeding; Renal Insufficiency, Chronic; Obesity
Keywords: time-restricted feeding; chronic kidney disease; obesity
MeSH Terms: conditions — Intermittent Fasting; Renal Insufficiency, Chronic; Obesity

STUDY DESIGN:
Intervention Model Description: It was non-randomized trial study design, two parallel groups were assigned to time-restricted feeding(TRF) and control group and to do the intervention for 12 weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-restricted feeding(TRF) (Experimental): The TRF group was asked to restrict the eating window to 8 hours a day, during waking hours and also continue a low-protein diet.
  Interventions: Behavioral: Time-restricted feeding(TRF)
- Control (No Intervention): The control group was asked to continue their usual low-protein diet eating schedule and pattern.

INTERVENTIONS:
Behavioral: Time-restricted feeding(TRF) — The TRF group was asked to restrict the eating window to 8 hours a day, during waking hours and also continue a low-protein diet.
  Arms: Time-restricted feeding(TRF)

SUMMARY:
Obesity is associated with glomerular hyperfiltration leading to renal impairment and is a risk factor for the progression of kidney disease.Weight loss can reduce proteinuria and improve eGFR.Intermittent fasting is safe and effective, and in addition to improving body shape and weight in obese patients, it can also improve glucolipid metabolism, reduce proteinuria, improve kidney function and delay the progression of kidney disease.

DETAILED DESCRIPTION:
KDOQI clinical practice guideline for nutrition in chronic kidney disease (CKD) uses a low-protein diet to reduce renal impairment and delay progression. The current research hotspot is dietary intervention. Time-restricted feeding was used to intervene in the progression of CKD. It restrict the time of eating but not the eaten calories, which have a higher compliance and safety. Studies have shown that intermittent fasting in obese patients with CKD is not only reduce body weight, but also improves glycolipid metabolism, reduces proteinuria and delays the progression of kidney disease. Intermittent fasting is currently a scientific research hotspot, and there are few international studies on the implementation of intermittent fasting to delay the deterioration of renal function in obese CKD patients, and lack of data on Chinese patients, which has great research potential. Based on the above background, this study was conducted as an pilot clinical trial to explore the effects of intermittent fasting on obese patients with CKD and to observe its effectiveness, safety and compliance.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* CKD stage 3-4 and not on dialysis (eGFR: 15-59ml/min/1.73m2)
* BMI ≥ 25 kg/m2
* Good reading and comprehension skills, simple smartphone operation and no communication difficulties
* Signed informed consent

Exclusion Criteria:

* Pregnant and breastfeeding
* End-stage diseases
* Acute and active diseases such as gastrointestinal bleeding or acute infections, serious decompensation with diseases such as cirrhosis decompensation stage, malignant tumor, serious heart and lung diseases, severe primary diseases of hematopoietic system, severe hypertension (systolic blood pressure ≥200mmHg, diastolic blood pressure ≥120mmHg) and difficult to control blood pressure, within 3 months after major surgery, such as open surgery
* Mental patients
* Using medium-high doses of hormones and immunosuppressants
* Participating in other researchers
* Taking other dietary therapies, undergoing weight loss treatment
* Vegetarian
* Type 1 diabetes and type 2 diabetes using insulin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Change in eGFR (ml/min/1.73m2) | 12 weeks
  eGFR at final visit - eGFR at initial visit

SECONDARY OUTCOMES:
Changes in body weight (Kilograms) | 12 weeks
  body weight at final visit - body weight at initial visit
Changes in waist circumference (cm) | 12 weeks
  waist circumference at final visit - waist circumference at initial visit
Change in body mass index (kg/m2) | 12 weeks
  body mass index at final visit - body mass index at initial visit
Changes in serum total cholesterol levels (mmol/L) | 12 weeks
  serum total cholesterol levels at final visit - serum total cholesterol levels at initial visit
Changes in serum low density lipoprotein cholesterol levels (mmol/L) | 12 weeks
  serum low density lipoprotein cholesterol levels at final visit - serum low density lipoprotein cholesterol levels at initial visit
Changes in serum triglyceride levels (mmol/L) | 12 weeks
  serum triglyceride levels at final visit - serum triglyceride levels at initial visit
Changes in serum high density lipoprotein cholesterol levels (mmol/L) | 12 weeks
  serum high density lipoprotein cholesterol levels at final visit - serum high density lipoprotein cholesterol levels at initial visit
Changes in serum albumin (g/L) | 12 weeks
  serum albumin at final visit - serum albumin at initial visit
Changes in total serum protein (g/L) | 12 weeks
  total serum protein at final visit - total serum protein at initial visit
Changes in fat free mass (kg) | 12 weeks
  fat free mass at final visit - fat free mass at initial visit
Changes in body fat mass (kg) | 12 weeks
  body fat mass at final visit - body fat mass at initial visit
Changes in percent body fat (%) | 12 weeks
  percent body fat at final visit - percent body fat at initial visit
Changes in waist-hip ratio | 12 weeks
  waist-hip ratio at final visit - waist-hip ratio at initial visit
Changes in soft lean mass (kg) | 12 weeks
  soft lean mass at final visit - soft lean mass at initial visit
Changes in visceral fat area (cm2) | 12 weeks
  visceral fat area at final visit - visceral fat area at initial visit
Changes in arm circumference (cm) | 12 weeks
  arm circumference at final visit - arm circumference at initial visit
Changes in triceps skin fold thickness (cm) | 12 weeks
  triceps skin fold thickness at final visit - triceps skin fold thickness at initial visit
Changes in grip strength (kg) | 12 weeks
  grip strength at final visit - grip strength at initial visit
Changes in fasting blood glucose (mmol/L) | 12 weeks
  fasting blood glucose at final visit - fasting blood glucose at initial visit
Changes in serum creatinine (umol/L) | 12 weeks
  serum creatinine at final visit - serum creatinine at initial visit
Changes in blood urea nitrogen (mmol/L) | 12 weeks
  blood urea nitrogen at final visit - blood urea nitrogen at initial visit
Changes in serum uric acid (umol/L) | 12 weeks
  serum uric acid at final visit - serum uric acid at initial visit
Changes in proteinuria creatinine ratio (g/g) | 12 weeks
  proteinuria creatinine ratio at final visit - proteinuria creatinine ratio at initial visit
Changes in serum cystatin C (mg/L) | 12 weeks
  serum cystatin C at final visit - serum cystatin C at initial visit
Changes in total urine urea in 24 hours (mmol/24h) | 12 weeks
  total urine urea in 24 hours at final visit - total urine urea in 24 hours at initial visit
Changes in interleukin-6 (pg/mL) | 12 weeks
  interleukin-6 at final visit - interleukin-6 at initial visit
Changes in tumor necrosis factor-α (pg/mL) | 12 weeks
  tumor necrosis factor-α at final visit - tumor necrosis factor-α at initial visit
Changes in C-reactive protein (mg/L) | 12 weeks
  C-reactive protein at final visit - C-reactive protein at initial visit
Changes in species of intestinal flora | 12 weeks
  species of intestinal flora at final visit - species of intestinal flora at initial visit

OTHER OUTCOMES:
Changes in hunger scores | Weeks 6 and 12
  Assessed using Visual Analog Scales (VAS with a scale of 1-10)
Changes in fatigue scores | Weeks 6 and 12
  Assessed using Visual Analog Scales (VAS with a scale of 1-10)
Changes in satiety scores | Weeks 6 and 12
  Assessed using Visual Analog Scales (VAS with a scale of 1-10)
Changes in gastrointestinal flatulence scores | Weeks 6 and 12
  Assessed using Visual Analog Scales (VAS with a scale of 1-10)
Changes in nausea and vomiting scores | Weeks 6 and 12
  Assessed using Visual Analog Scales (VAS with a scale of 1-10)
Changes in constipation scores | Weeks 6 and 12
  Assessed using Visual Analog Scales (VAS with a scale of 1-10)
Changes in diarrhea scores | Weeks 6 and 12
  Assessed using Visual Analog Scales (VAS with a scale of 1-10)
Changes in dry mouth and bitterness scores | Weeks 6 and 12
  Assessed using Visual Analog Scales (VAS with a scale of 1-10)
Changes in dizziness and headache scores | Weeks 6 and 12
  Assessed using Visual Analog Scales (VAS with a scale of 1-10)
Changes in irritability scores | Weeks 6 and 12
  Assessed using Visual Analog Scales (VAS with a scale of 1-10)
Changes in anxiety scores | Weeks 6 and 12
  Assessed using Visual Analog Scales (VAS with a scale of 1-10)
Changes in depression scores | Weeks 6 and 12
  Assessed using Visual Analog Scales (VAS with a scale of 1-10)

CONTACTS AND LOCATIONS:
Overall Officials: Xu-sheng Liu, M.M, Study Chair — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No